CLINICAL TRIAL: NCT00734448
Title: Effect of Myo-inositol Administration on Insulin Sensitivity in Gestational Diabetes Patients by Continuous Glucose Monitoring System (CGMS)
Brief Title: Myo-inositol Administration in Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Rosario D'anna, associate professor, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Myo-1954
Record Dates: First submitted 2008-04-16; First posted 2008-08-14 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Gestational Diabetes Mellitus
Keywords: gestational diabetes mellitus; carbohydrate intolerance; myo-inositol; insulin resistance
MeSH Terms: conditions — Diabetes, Gestational; Glucose-Galactose Malabsorption; Insulin Resistance | interventions — Inositol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A,1 (Experimental): Gestational diabetes patients who take myo-inositol
  Interventions: Dietary Supplement: myo-inositol

INTERVENTIONS:
Dietary Supplement: myo-inositol — 2 g twice a day until delivery

SUMMARY:
Myo-Inositol is an insulin sensitizing agent that ameliorate the insulin resistance in women affected by gestational diabetes (GDM), but there is no information about the effect on the glucose profile. Maternal hyperglycemia of GDM, especially hypoglycemic excursions, are associated with adverse pregnancy outcome. Continuous Glucose Monitoring System (CGMS) is obviously better than intermittent self monitoring in detecting glucose profile and magnitude and duration of glucose fluctuations. For this reason, we propose a clinical trial to analyze the characteristics of glucose variability in GDM women,treated with diet and folic acid alone or with diet, folic acid and myo-inositol supplementation.

DETAILED DESCRIPTION:
Our study is a randomized, prospective, controlled trial, including the first 30 consecutive Caucasian gestational diabetes patients diagnosed,according the International Association of Diabetes and Pregnancy Study Group (IADPSG) panel criteria, from November 2013 in the Department of Obstetric and Gynecology of Messina University (ITALY). After an informed consent they will be randomly assigned to receive (n. 15) diet and folic acid (400 mcg per day) alone or (n. 15) diet, folic acid (400 mcg per day) and myo-inositol (2 g. twice a day)supplementation. The insulin sensitivity index (HOMA-IR) and the glycemic profile will be monitor by CGMS for each patient at GDM diagnosis and after 8 weeks of treatment The pregnant women who will delivery before the time treatment (8 weeks) or who need insulin will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Gestational diabetes diagnosed within 28 weeks
* Caucasian pregnant women

Exclusion Criteria:

* Non Caucasian pregnant women
* Delivery before 8 weeks of treatment

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity index (HOMA-IR) and continuous glucose monitoring profile | Change from baseline in HOMA-IR at 8 weeks of treatment

SECONDARY OUTCOMES:
baby weight at delivery | After delivery

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, professor, Principal Investigator — University of Messina, ITALY
Locations (1):
- University of Messina -, Messina, Sicily, Italy